CLINICAL TRIAL: NCT00866762
Title: A Phase II Study of MK-0683 in Patients With Polycythaemia Vera and Essential Thrombocythaemia.
Brief Title: A Study of the Efficacy of MK-0683 in Patients With Polycythaemia Vera and Essential Thrombocythaemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-0683/092-0
Record Dates: First submitted 2009-03-17; First posted 2009-03-20 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
Keywords: Polycythaemia Vera; Polycythemia Vera; Essential Thrombocythaemia; Essential Thrombocythemia; HDAC-inhibitor; Haematology; Hematology; Haematological disorder; Haematological disease; Hematological disorder; Hematological disease
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Polycythemia; Hematologic Diseases | interventions — Histone Deacetylase Inhibitors; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment with study drug approximately 6 months and follow-up for 3 months
  Interventions: Drug: HDAC inhibitor (MK-0683)

INTERVENTIONS:
Drug: HDAC inhibitor (MK-0683) — 400 mg once daily for 6 months

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of MK-0683 in the treatment of PV and ET. This agent has most recently been shown to be a potent inhibitor of the autonomous proliferation of haematopoietic cells of PV and ET patients carrying the JAK2 V617F mutation. Accordingly, it may be anticipated that MK-0683 - by decreasing the JAK2 allele burden - may influence clonal myeloproliferation and in vivo granulocyte, platelet and endothelial activation , which are considered to be major determinants of morbidity and mortality ( thrombosis, bleeding, extramedullary haematopoiesis , myelofibrosis ) in these disorders. The effects of MK-0683 at the molecular level will be studied by global/ focused gene expression profiling, epigenome profiling and proteomics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient > 18 years of age AND
* A confirmed diagnosis of PV AND
* Biochemical evidence of active disease as defined by:

  * a need for phlebotomy within last 3 months
  * a leukocyte count > 10 x 10^9/L in the absence of infection or inflammation (normal CRP) and/or (PV/ET)
  * a platelet count > 450 x 10^9/L in the absence of infection or inflammation (normal CRP)(PV/ET) OR
* Male or female patient > 18 years of age AND
* A confirmed diagnosis of ET AND
* Biochemical evidence of active disease as defined by *a platelet count > 450 x 10^9/L in the absence of infection or inflammation

Inclusion Criteria for both PV and ET:

* Newly diagnosed or previously treated patient in chronic phase OR
* Advanced phase PV or ET as defined by blasts of > 1 x 10^9/L in the peripheral blood and/or white cell count > 30 x 10^9/L OR
* Resistant or refractory PV or ET as defined by haemoglobin < 10.5 gm/dl with a platelet count > 600 x 10^9/L on current therapy OR
* Cycling platelet counts on therapy OR
* Intolerant to other therapies defined by patients with PV or ET who have side effects on current therapies preventing continuation (leg ulcers on hydroxycarbamide, unacceptable fatigue etc on interferon)

Exclusion Criteria:

* A platelet count > 1500 x 10^9/L (a need for cytoreduction in platelet count)
* Patients of childbearing potential without a negative pregnancy test prior to initiation of study drug
* Women who are breast feeding
* Males and females not using contraceptives if sexually active.
* EGOC Performance status Score > or = 3
* Serum creatinine more than 2 x's teh ULN
* Total serum bilirubin more than 1.5 x's the ULN
* Serum AST/ALT more than 3 x's the ULN
* Interferon alpha within 1 week of day 1
* Hydroxycarbamide within 1 week of day 1
* Anagrelide within 1 week of day 1
* Valproic acid (as an anticonvulsant) within 28 days of day 1
* Any other investigational drug within 28 days of day 1
* Active HIV, HBV or HCV infection
* Any serious concomitant disease or circumstances that could limit compliance with the study, including but not limited to the following: CTCAE grade 3-4 cardiac general & arrhythmia, or psychiatric or social conditions that may interfere with patient compliance.
* Any prior malignancy with the exception of cervical intraepithelial neoplasia, basal cell carcinoma of the skin, or other localized malignancy that has undergone potentially curative therapy with no evidence of that disease for five years, and who is deemed to be at low risk for recurrence by his/her treating physician.
* Patient has a known allergy or hypersensitivity to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of study drug (MK-0683) in the treatment of patients with PV and ET. | one year

SECONDARY OUTCOMES:
To study changes in bone marrow morphology before and after treatment with study drug. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Hasselbalch, MD, Principal Investigator — Department of Hematology, Copenhagen University Hospital Herlev
Locations (16):
- Denmark (6):
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Esberg Hospital, Esbjerg
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Regional Hospital Viborg, Viborg
- VU University Medical Centre, Amsterdam, Netherlands
- Sweden (5):
  - University Hospital Orebro, Örebro
  - Stockholm South General Hospital (Sodersjukhuset), Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
  - Sahlgrenska University Hospital & Uddevalla Hospital, Uddevalla
  - Uppsala University Hospital, Uppsala
- United Kingdom (4):
  - Centre for Cancer Research and Cell Biology, Queen's University Belfast, Belfast, Northern Ireland
  - Cardiff University, Cardiff
  - Russell's Hall Hospital, Dudley
  - St Thomas' Hospital, London